CLINICAL TRIAL: NCT05295186
Title: Noninvasive Assessment of Respiratory Mechanics, Inspiratory Effort, and Respiratory Drive During Spontaneous Breathing Trial to Predict Extubation Failure in High-Risk Patients
Brief Title: Non-invasive Respiratory Monitoring During SBT
Status: Completed | Type: Observational
Sponsor: University of Bari (Other)
Collaborators: Università degli Studi di Ferrara (Other); Catholic University of the Sacred Heart (Other); Università degli Studi di Sassari (Other); University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Salvatore Grasso, PROF, University of Bari
Other Study IDs: SBT_PAV01
Record Dates: First submitted 2022-03-09; First posted 2022-03-25 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2024-04

CONDITIONS: Mechanical Ventilation Complication; Acute Respiratory Failure; Re-intubation Rate
Keywords: spontaneous breathing trial; Extubation failure; lung mechanics; airway occlusion pressure; noninvasive monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients at high-risk for re-intubation

SUMMARY:
Spontaneous breathing trials (SBTs) assess readiness for extubation, yet the use of conventional parameters used to establish weaning success may be elusive, especially in high-risk patients. Currently, non-invasive techniques allow comprehensive bedside assessment of advanced respiratory mechanics, including metrics of respiratory system compliance (CRS), respiratory muscle effort (POCC) and respiratory drive intensity (P0.1). This study investigates whether these measurements during SBT may improve the prediction of extubation outcomes

ELIGIBILITY:
To be eligible, patients had to meet all of the following criteria:

1. Age ≥ 18 years.
2. The presence of ≥ 1 among the following factors to define the high-risk for re-intubation: age older than 65 years; heart failure as the primary indication for mechanical ventilation; moderate to severe chronic obstructive pulmonary disease (COPD); an Acute Physiology and Chronic Health Evaluation II (APACHE II) score higher than 12 on extubation day; body mass index of more than 30; inadequate cough reflex or suctioning >2 times within 8 hours before extubation; prolonged use of invasive ventilation (≥ 7 days from the first SBT); more than 2 comorbidities categorized based on the Charlson Comorbidity Index.
3. Deemed ready to be weaned from the ventilator, based on the following criteria: (a) invasive mechanical ventilation for more than 48 hours, including at least 12 hours of pressure support ventilation with PEEP ≤ 8 cmH2O and pressure support ≤ 10 cmH2O; (b) Improvement of the condition leading to intubation; (c) patient making inspiratory effort; (d) adequate gas exchange, as indicated by a ratio of partial pressure of arterial oxygen (PaO2) to inspiratory fraction of oxygen (FiO2) ≥ 150 with FiO2 ≤ 40% and arterial pH within normal range (7.30 - 7.50); (e) Glasgow Coma Score higher than 13; (f) a core temperature below 38°C; (g) Richmond agitation and sedation scale between -1 and +1.

Eligibility required readiness for scheduled extubation after successfully completing a 30-minute SBT in the pressure-support mode (7 cmH₂O)

SBT success was defined by the following criteria [19]: (a) adequate gas exchange, as indicated by a ratio of partial pressure of arterial oxygen (PaO2) to inspiratory fraction of oxygen (FiO2) ≥ 150 with FiO2 ≤ 40% and arterial pH within the normal range (7.30 - 7.50); (b) respiratory rate < 35/min; (c) spontaneous tidal volume higher than 5 ml of predicted body weight (PBW); (d) a ratio of respiratory rate to tidal volume (i.e. the rapid shallow breathing index, RSBI) < 105/min per liter; (e) systolic blood pressure between 90 and 160 mmHg and heart rate < 140/min, with or without low doses of vasopressors (< 0.5 mcg/kg/min). Exclusion criteria were tracheostomy, patients undergoing withdrawal of life-sustaining treatments, known neuromuscular diseases.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: High-risk patients for re-intubation were defined as follow :
  The presence of ≥ 1 among the following factors to define the high-risk for re-intubation: age older than 65 years; heart failure as the primary indication for mechanical ventilation; moderate to severe chronic obstructive pulmonary disease (COPD); an Acute Physiology and Chronic Health Evaluation II (APACHE II) score higher than 12 on extubation day; body mass index of more than 30; inadequate cough reflex or suctioning >2 times within 8 hours before extubation; prolonged use of invasive ventilation (≥ 7 days from the first SBT); more than 2 comorbidities categorized based on the Charlson Comorbidity Index.
Sampling Method: Probability Sample
Enrollment: 238 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Advance Respiratory mechanics assessment during SBT | 30 minutes
  The primary endpoint was to establish whether changes in CRS, POCC and P0.1 and/or their absolute values at the end of the PAV+ SBT differed between patients who subsequently required reintubation vs. those who were successfully extubated

SECONDARY OUTCOMES:
discriminatory power | 72 hours
  we aimed to test the discriminatory power of the absolute values of CRS, POCC and P0.1 at the end of SBT and discriminatory power of the SBT-induced percentage changes in these measurements during the trial in identifying patients who failed extubation.The decision to reintubate was made by the attending physicians, who were unaware of the study measurements results.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Azienda Ospedaliero Universitaria Policlinico, Bari
  - Salvatore Grasso, Bari

REFERENCES:
- [Derived] Murgolo F, Spadaro S, Grieco DL, Bertoni M, Pisani L, Spinazzola G, Di Mussi R, Michi T, Bartolomeo N, Fanelli V, Terragni P, Antonelli M, Ranieri VM, Grasso S. Assessment of Respiratory Mechanics and Inspiratory Effort During Spontaneous Breathing Trials to Predict Extubation Failure in High-Risk Patients. Am J Respir Crit Care Med. 2025 Dec;211(12):2340-2351. doi: 10.1164/rccm.202503-0544OC. PMID 41072398